CLINICAL TRIAL: NCT04541563
Title: Neurostimulation & Depression Study
Brief Title: Fisher Wallace Neurostimulation & Depression Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ProofPilot (Industry)
Collaborators: Fisher Wallace (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2518
Record Dates: First submitted 2020-08-14; First posted 2020-09-09 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: This is a fully remote trial where participants engage at home in the study using the ProofPilot study platform. All potential participant enrollment data, including proof of identity via government ID will be reviewed by licensed medical professionals in the participant's state prior to their full enrollment.
  Participants will be randomized into an immediate or delayed treatment arm. The immediate treatment arm participants will be shipped an active Fisher Wallace device limited to Level 2 output even if a participant raises the dial beyond that. The participant will remain with the active device for the full 8 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a fully remote trial. Participants will be randomized in ProofPilot, and only the fulfillment center will know whether the participant is in the placebo or control arm.
  Participants will be unblinded at week 4 at the crossover.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Immediate Treatment Arm (Experimental): The immediate treatment arm participants will be shipped an active Fisher Wallace device limited to Level 2 output even if a participant raises the dial beyond that. The participant will remain with the active device for the full 8 weeks.
  Interventions: Device: Fisher Wallace Cranial Electrotherapy Stimulator Device
- Delayed Treatment Arm (Sham Comparator): In the delayed treatment arm, the participants will receive a sham device that looks exactly the same, but only provides treatment for 2 seconds. At week 4, sham arm participants will be unblinded and shipped an active device (limited to Level 2 output even if a participant raises the dial beyond that). The delayed arm participants will continue with active devices for the remaining 4 weeks of the trial.
  Interventions: Device: Fisher Wallace Cranial Electrotherapy Stimulator Device

INTERVENTIONS:
Device: Fisher Wallace Cranial Electrotherapy Stimulator Device — Fisher Wallace Stimulator®, a patented cranial electrotherapy stimulation device that was cleared by the FDA in 1991 for the treatment of depression, anxiety and insomnia.

SUMMARY:
Examine the safety and effectiveness of the Fisher Wallace Cranial Electrotherapy Stimulator Device on Major Depressive Disorder using two 20-minute per day treatment sessions over eight weeks.

ELIGIBILITY:
Inclusion criteria:

* Age greater than or equal to 21
* US resident
* Can receive packages to their home via UPS/Fedex/USPS
* Major Depressive Disorder
* PHQ-8 Score greater than 10 (show some signs of mild to moderate depression)
* PHQ-8 Score less than 20 (given remote study serious depressed should be excluded)
* Read/write English
* have not contemplated suicide in the past year
* not been institutionalized for mental health issues.
* not currently experiencing problems with alcohol or drug abuse
* can commit to not drinking alcohol 4 hours before bedtime for the duration of the study
* can commit to two (2) 20 minute sessions per day for 8 weeks
* has not used a brain stimulation treatment in one year
* no suspected or known history of heart disease
* no pacemaker
* not under medical supervision for other serious medical condition
* not taking opioids
* is a resident of states in which we have licensed medical professionals

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Depression Inventory Score Baseline vs week 4 | Week 4
  Change in depression symptoms from baseline to treatment week 4 in immediate versus delayed arm. Lower scores show improvement in depression symptoms.

SECONDARY OUTCOMES:
Systematic Assessment for Treatment Emergent Events (SAFTEE) at week 8 | Week 8
  assessment at week tolerability, safety and adherence at week 8
Change in Patient Health Questionnaire - 8 (PHQ-8) Score Baseline vs week 4 | Week 4
  Change in self reported depression self assessed at baseline and week 4. Lower scores in the PHQ-8 show improvement in depression symptoms
Change in Patient Health Questionnaire - 8 (PHQ-8) Score Baseline vs week 2 | Week 2
  Change in self reported depression self assessed at baseline and week 2. Lower scores in the PHQ-8 show improvement in depression symptoms.
Change in Beck Depression Inventory Score Delay Arm Week 4 to Week 8 | Week 8
  Participants will self assess at point of receiving active device at crossover for the remaining 4 weeks of the trial. Lower scores show improvement in depression symptoms.
Change in Hamilton Depression Score Baseline vs week 4 | Week 4
  Participants will be assessed by a tele-psychiatrist at baseline and week 4. Lower scores show improvement in depression symptoms.
Change in Hamilton Depression Score Baseline vs week 2 | Week 2
  Participants will be assessed by a tele-psychiatrist at baseline and week 2. Lower scores show improvement in depression symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- ProofPilot (Remote Virtual Trial), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT04541563/Prot_000.pdf
  • Informed Consent Form (2020-08-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT04541563/ICF_001.pdf